CLINICAL TRIAL: NCT04090944
Title: Comparison Between Blind And Ultrasound Guided Laryngeal Mask Airway Insertion In Adult Patients Undergoing Elective Surgery: A Randomized Control Study
Brief Title: Comparison Between Blind And Ultrasound Guided Laryngeal Mask Airway Insertion
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, mohammed abd elrehman moselhy, Mohammed Abd Elrehman Moselhy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Beni-suef Hospital
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: the Position of Laryngeal Mask Airway

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st group (group B) (Active Comparator): The LMA LarySeal Multiple will be inserted using the blind technique which involves holding the LMA like a pen guided into the pharynx with the index finger of the operator at the junction of the tube and the bowl, with the operator at the head of the patient and the LMA facing caudally.
  The position of LMA will be assessed by another anesthetist (blinded assessor) using the fiberoptic laryngoscope (KARL STORZ 11301BN1, Germany) per the grading devised by Aoyama et al.
  Interventions: Procedure: the fiberoptic laryngoscope (KARL STORZ 11301BN1, Germany) for confirmation of LMA position
- 2nd group:(group U) (Active Comparator): The LMA LarySeal Multiple will be inserted under the guide of B-mode US on the anterior neck . Transverse scans , Sagittal view and Parasagittal view.
  -The position of LMA will be assessed by another anesthetist (blinded assessor) using the fiberoptic laryngoscope (KARL STORZ 11301BN1, Germany) per the grading devised by Aoyama et al.
  Interventions: Procedure: the fiberoptic laryngoscope (KARL STORZ 11301BN1, Germany) for confirmation of LMA position

INTERVENTIONS:
Procedure: the fiberoptic laryngoscope (KARL STORZ 11301BN1, Germany) for confirmation of LMA position — -The position of LMA will be assessed by another anesthetist (blinded assessor) using the fiberoptic laryngoscope (KARL STORZ 11301BN1, Germany) per the grading licensed by Aoyama et al.

SUMMARY:
The Proper position of a laryngeal mask airway (LMA) requires confirmation to ensure the adequacy of laryngeal seal and pulmonary ventilation. This confirmation may help in prevention of the peri-operative airway complication and ventilation events associated with LMA placement

DETAILED DESCRIPTION:
It is common practice to inflate the cuff of LMA with the maximum recommended volume (size 3, 20 ml; size 4, 30 ml; size 5, 40 ml), as illustrated in several studies , but it may become more rigid which may cause displacement of the LMA and decreases the airway sealing of LMA, more pressure on pharyngeal mucosa which might cause severe mucosal ischemia leading to post- operative sore throat, dysphagia or hoarseness.

Ultrasonography can reliably confirm correct placement of supraglottic devices like laryngeal mask airway (LMA) and rules out causes of inadequate ventilation , also it was found to be a sensitive in detecting rotational malposition of LMA in children.

the replacement of air with saline in LMA cuffs enable detection of cuffs in the airway allowing visualization of the surrounding structures and tissues as the ultrasound beam can be transmitted through the fluid-filled cuffs without being reflected from air mucosal interface.

the adequacy of LMA position will be confirmed by a fiberoptic laryngoscope (FOL)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18- 60 years of either sex, ASA physical status I - II, weighting 50-100 kg, who will scheduled for elective surgery under general anesthesia.

Exclusion Criteria:

* - Patients whom LMA is contraindicated as patients who are at an increased risk of gastric aspiration as (obstetrics, hiatal hernia or esophageal reflux ), patients with high airway resistance e.g. (bronchospasm or pulmonary edema), patients with low pulmonary compliance e.g. (obesity), cases of an inability to open the mouth or an infection or pathologic abnormality within the oral cavity or pharynx and nonsupine position of operation .
* Patients with a known or predicted difficult airway as patients with class III and IV Modified Mallampati Score or with score > 5 wilson's risk score.
* Patients with cardiovascular disease (congestive heart failure, coronary artery disease), history of renal or hepatic insufficiency, and endocrinal Diseases will be excluded from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
the Score of the fibreoptic view of the larynx | from the clinical judgement of correct position (as ventilation without substantial leak at an airway pressure ≤20 cm H2O, observation of EtCO2 trace )up to 120 second
  the aim of this study is to compare between the blind technique and US guided technique of laryngeal mask airway insertion regarding the position as confirmed by the fiberoptic laryngoscope.

CONTACTS AND LOCATIONS:
Overall Officials: mohammed abd moselhy, MD, Principal Investigator — lecturer in anesthesia
Locations (1):
- Beni-suef University Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No